CLINICAL TRIAL: NCT02138383
Title: A Phase I Trial With Cohort Expansion of Enzalutamide in Combination With Gemcitabine and Nab-Paclitaxel for the Treatment of Advanced Pancreatic Cancer
Brief Title: Enzalutamide in Combination With Gemcitabine and Nab-Paclitaxel for the Treatment of Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17696
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Cancer
Keywords: advanced pancreatic cancer; pancreas; malignant neoplasm; endocrine system
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — enzalutamide; Receptors, Androgen; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Tubulin Modulators

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation and Dose Expansion (Experimental): Dose Escalation: To find the dose of enzalutamide that can be safely given with gemcitabine and nab-paclitaxel in patients with advanced pancreatic cancer.
  Dose Expansion: To find the effect on tumor of the combination of enzalutamide, gemcitabine and nab-paclitaxel.
  Interventions: Drug: Enzalutamide; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Enzalutamide — The starting dose of enzalutamide will be 80 mg (Level 1) daily, taken orally. The dose escalation schedule is a standard 3 + 3 design. In the first part of the study, different doses of enzalutamide will be tested. In the second part of the study, all patients will be started at the same dose of enzalutamide.
  Other Names: MDV3100; XTANDI®; androgen receptor (AR) antagonist
Drug: Gemcitabine — The starting dose of gemcitabine will be 1000 mg/m^2 administered intravenously on days 1, 8 and 15 of each cycle.
  Other Names: nucleoside inhibitor; GEMZAR®
Drug: Nab-paclitaxel — The starting dose of nab-paclitaxel will be 125 mg/m^2 administered intravenously on days 1, 8 and 15 of each cycle.
  Other Names: albumin bound paclitaxel; microtubule inhibitor; Abraxane®

SUMMARY:
The main purpose of this study is to find out the dose of enzalutamide that can be safely given with gemcitabine and nab-paclitaxel in patients with advanced pancreatic cancer. Researchers also want to find out the side effects of these drugs when given together. This study will help in finding out the effect on tumor of the combination of enzalutamide, gemcitabine and nab-paclitaxel. In the first part of the study, different doses of enzalutamide will be tested. In the second part of the study, all patients will be started at the same dose of enzalutamide.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed pancreatic adenocarcinoma that is metastatic or unresectable. In the dose expansion phase, the tumor must express Androgen Receptor (AR) by immunohistochemistry. If ≥1% of the tumor cells express AR, it will be considered positive for this trial.
* Must have measurable disease per Response Criteria in Solid Tumors (RECIST) criteria version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status <2 (Karnofsky >60%)
* Life expectancy of greater than 3 months
* Must have normal organ and marrow function
* Prior treatment with gemcitabine alone or 5-Fluorouracil with radiation as an adjuvant therapy will be allowed; Should not have received gemcitabine within 6 months of starting the study treatment; 5-Fluorouracil or radiation treatment should be received more than 4 weeks prior to receiving the study drug.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of the study treatment.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Prior treatment with any cytotoxic chemotherapy except as an adjuvant therapy. Participant should not have received gemcitabine within 6 months of starting the study treatment. 5-Fluorouracil or radiation treatment should be received more than 4 weeks prior to receiving the study drug.
* May not be receiving any other investigational agents within 4 weeks of starting the study treatment and during the study period.
* Untreated brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, nab-paclitaxel or enzalutamide.
* Have undergone major surgery within 4 weeks prior to starting the study treatment.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements; history of myocardial infarction within 6 months of starting study treatment.
* Known history of human immunodeficiency virus (HIV) infection or active hepatitis B or hepatitis C
* Any history of seizure. History of loss of consciousness or transient ischemic attack within 12 months of starting the study drug.
* Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control
* Chronic treatment with immunosuppressant drugs
* Other malignancy requiring active treatment
* Any significant medical condition, laboratory abnormality, or psychiatric illness, that would prevent participating in the study, including the inability to swallow capsules
* Any active infection not controlled by antibiotics
* Concomitant medications that lower seizure threshold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-05-22 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2019-10-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Up to 18 months
  To determine the maximally tolerated dose (MTD) of enzalutamide in combination with gemcitabine and nab-paclitaxel in advanced pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States